CLINICAL TRIAL: NCT01284959
Title: Different Safety Profile of Risperidone and Paliperidone Extended-release: a Double-blind, Placebo-controlled Trial With Healthy Volunteers
Brief Title: Different Safety Profile of Risperidone and Paliperidone Extended-release
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: AstraZeneca (Industry); Janssen Korea, Ltd., Korea (Industry); Korea Otsuka Pharmaceutical Co., Ltd. (Industry); Sanofi-Synthelabo (Industry)
Responsible Party: Principal Investigator, Young Chul Chung, Professor of Psychiatry, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CBIRB1005-58
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia
Keywords: cognitive function; subjective experiences; neuroleptic-induced deficit syndrome; paliperidone extended-release; risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- risperidone (Experimental): Drug: risperidone 3mg, PO two times Groups: risperidone
  Interventions: Drug: risperidone
- placebo (Placebo Comparator): drug: lactose, PO 3 times group: placebo
  Interventions: Drug: placebo
- paliperidone ER (Experimental): drug : Paliperidone ER 6mg PO, two times group: paliperidone ER
  Interventions: Drug: paliperidone ER

INTERVENTIONS:
Drug: risperidone — risperidone 3mg, PO, 3 times
  Other Names: Rispedal
  Arms: risperidone
Drug: paliperidone ER — paliperidone ER 6mg, PO,3 times
  Other Names: Invega
  Arms: paliperidone ER
Drug: placebo — lactose PO, 3times
  Arms: placebo

SUMMARY:
The main objective of this study was to assess subjective experiences related to secondary negative symptoms and cognitive performance in healthy volunteers in response to multiple doses of paliperidone ER and risperidone in a double-blind, placebo-controlled trial. Adverse events caused by these drugs were also evaluated.

DETAILED DESCRIPTION:
A new oral antipsychotic drug, paliperidone extended-release (ER), has recently been developed and might represent an innovative approach in the treatment of schizophrenia. Paliperidone is 9-hydroxyrisperidone, the chief active metabolite of risperidone. Although paliperidone possesses a pharmacological profile very similar to that of its parent compound, it has many different pharmacokinetic and pharmacodynamic characteristics compared with risperidone (Pani and Marchese, 2009). First, paliperidone ER utilizes an osmotic controlled-release oral delivery system (OROS), resulting in a more stable serum concentration and reduced likelihood of causing unexpected over- or under-dosages due to CYP2D6 genetic variability. Second, paliperidone does not undergo significant hepatic metabolism, and the drug is predominantly excreted by the kidney as an unchanged drug; whereas risperidone is extensively metabolized by the CYP2D6 hepatic enzyme. Third, the off-rate for dissociation from human cloned D2 receptors in tissue culture cells is faster for paliperidone (60 s) compared with risperidone (27 min) (Seeman, 2005). Due to its looser binding to D2 receptors, paliperidone should be associated with a reduced risk of extrapyramidal side effects compared with its parent drug. Fourth, ex vivo studies have indicated that paliperidone injections induce relatively smaller H1 occupancy levels in the brains of animals when compared with similar dosages of risperidone (Schotte, et al. 1995 and 1996). This may contribute to a reduced sedative effect and less weight gain secondary to paliperidone when compared with risperidone. Finally, paliperidone has no relevant affinity toward muscarinic receptors, resulting in the absence of anticholinergic side effects; this is another important benefit compared with risperidone (Schotte, et al. 1996). Therefore, paliperidone would be the drug of choice in young psychotic patients for whom preservation or improvement of cognitive function is critical. All of these properties might be associated with improved efficacy and better tolerability of paliperidone ER compared with risperidone. In support of this view, recent studies (Canuso, et al. 2008 and 2010) demonstrated that switching from risperidone to paliperidone ER resulted in improvements in medication satisfaction, Positive and Negative Syndrome Scale (PANSS) (Kay, et al. 1987) score, and abbreviated Extrapyramidal Symptoms Rating Scale (Chouinard and Margolese, 2005) score. However, to date, no clinical trials have investigated the relative superiority of paliperidone ER over risperidone in terms of effects on cognitive function. Recently, interest in the negative subjective experiences secondary to antipsychotic medications has been renewed, as these experiences are key factors in adherence and clinical outcomes (Awad, 1993; van Putten and May, 1978). Artaloytia et al. (2006) reported that risperidone induced negative symptoms in healthy volunteers, which might be termed secondary negative symptoms. Therefore, we hypothesized that paliperidone ER has a better safety profile in terms of subjective experiences and cognitive function compared with risperidone. Research on the effects of antipsychotic drugs on subjective experiences and cognitive function in patients with schizophrenia may be hampered by numerous confounding factors, such as pathological features of the illness, patient motivation, or concomitant medications. Investigating the effects of antipsychotic drugs in healthy subjects provides a method for controlling these variables. Therefore, the main objective of this study was to assess subjective experiences related to secondary negative symptoms and cognitive performance in healthy volunteers in response to multiple doses of paliperidone ER and risperidone in a double-blind, placebo-controlled trial. Adverse events caused by these drugs were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-38 years and meet no DSM-IV diagnostic criteria as assessed by using the Structured Clinical Interview for DSM-IV, research version

Exclusion Criteria:

Anyone who:

* Participated in other clinical trials within 30 days from the start of this clinical trial or is currently participating in one
* Has progressive disease or in unstable medical condition unfit for the trial
* Has been diagnosed in psychiatric terms in the past, depends on psychotropic substance, or has overdosed or depended on the substance or alcohol (except for coffee or tobacco) within 1 month from the trial start
* Is suicidal or highly probable of suicides; OR
* Has test results considered clinically meaningful

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young-chul Chung, M.D., Ph.D., Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk national university hospital, Jeonju, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone: Drug: risperidone Groups: risperidone
- Placebo: drug: lactose group: placebo
- Paliperidone ER: Drug: Paliperidone ER Groups: Paliperidone ER
Period: Overall Study
Arm/Group | Risperidone | Placebo | Paliperidone ER
Started | 11 | 12 | 11
Completed | 10 | 12 | 10
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone | Placebo | Paliperidone ER | Total
Number analyzed (Participants) | 11 | 12 | 11 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 11 | 34
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.40 (2.59) | 28.08 (2.23) | 30.60 (3.27) | 28.97 (2.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 5 | 17
  Male | 4 | 7 | 6 | 17
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 11 | 12 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Negative Symptoms and Neuroleptic Induced Deficit Syndromes by Objective Rating Scales
Description: SANS(Scale for the Assessment of Negative Symptoms), NIDSS(Neuroleptic induced Deficit Syndrome Scale) In NIDSS, the average of number 1 to 5 is blunted affect, the average of number 16 to 20 is avolition, the average of number 6 to 15 is cognition, the average of all score is total.
  Minimum of NIDSS(avolition, blunted affect, cognition, total) is -3, maximum is +3.(subscale score and total) '+' is better outcome, '-' is worse outcome. Minimum of SANS-Global score for alogia and blunted affect is 0, Maximum of SANS-Global score for alogia and blunted affect is 5 The higher number is worse outcome. The zeros are measured and Calcuated value This outcome measure is reporting a change between baseline and 2hr after third medication.
Time Frame: baseline and 2hr after third medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Placebo | Paliperidone ER
Number analyzed (Participants) | 10 | 12 | 10
units on a scale
  NIDSS-Avolition | -1.30 (1.22) | -0.28 (0.64) | -0.66 (0.53)
  NIDSS-Blunted Affect | -0.70 (0.74) | 0.02 (0.35) | -0.24 (0.64)
  NIDSS-Cognition | -0.54 (0.53) | 0.02 (0.26) | -0.38 (0.39)
  NIDSS-Total | -0.77 (0.70) | -0.06 (0.35) | -0.42 (0.38)
  SANS-Global score for alogia | 0.67 (0.50) | 0 (0) | 0 (0)
  SANS-Global score for blunted affect | 0.67 (0.50) | 0 (0) | 0.10 (0.32)

2. Secondary Outcome: Assessment of Adverse Events by Objective Rating Scales and Self Report Scales
Description: DIEPSS(Drug-Induced Extrapyramidal Symptoms Scale), VAS(Visual analog scale);mental sedation (alert-drowsy, muzzy-clear headed, mentally slow-quick witted, attentive-dreamy), physical sedation (strong-feeble, well coordinated-clumsy, lethargic-energetic, incompetent-proficient), tranquilization (calm-excited, contented-discontented, troubled-tranquil, tense-relaxed), and other types of feelings (happy-sad, antagonistic-amicable, interested-bored, withdrawn-gregarious) Minimum of VAS(Mental sedation score,Physical sedation score,Total score) is 0, Maximum is 10.
  VAS-total score is average of all subscale scores. Minimum of DIEPSS is 0, Maximum is 4. The higher number is worse outcome. The score ranges are for subscale score. This outcome measure is reporting a change between baseline and 2hr after third medication.
Time Frame: baseline and 2hr after third medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Placebo | Paliperidone ER
Number analyzed (Participants) | 10 | 12 | 10
units on a scale
  VAS-Total score | 5.41 (1.82) | 3.35 (1.69) | 4.11 (1.63)
  VAS-Mental sedation score | 6.05 (2.14) | 3.85 (1.82) | 4.78 (1.56)
  VAS-Physical sedation score | 5.78 (1.79) | 3.23 (1.66) | 4.08 (1.94)
  DIEPSS-Bradykinesia score | 0.60 (0.52) | 0.08 (0.29) | 0.20 (0.42)

3. Secondary Outcome: Assessment of Adverse Events by Objective Rating Scales and Self Report Scales
Description: DIEPSS(Drug-Induced Extrapyramidal Symptoms Scale), VAS(Visual analog scale);mental sedation (alert-drowsy, muzzy-clear headed, mentally slow-quick witted, attentive-dreamy), physical sedation (strong-feeble, well coordinated-clumsy, lethargic-energetic, incompetent-proficient), tranquilization (calm-excited, contented-discontented, troubled-tranquil, tense-relaxed), and other types of feelings (happy-sad, antagonistic-amicable, interested-bored, withdrawn-gregarious) Minimum of VAS is 0, Maximum is 10 Minimum of DIEPSS is 0, Maximum is 4 The higher number is worse outcome. The score ranges are for subscale score. This outcome measure is reporting a change between baseline and 50hr after third medication.
Time Frame: baseline and 50hr after third medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Placebo | Paliperidone ER
Number analyzed (Participants) | 10 | 12 | 10
units on a scale
  VAS-Total score | 6.15 (1.27) | 3.74 (1.80) | 3.42 (1.75)
  VAS-Mental sedation score | 6.53 (1.37) | 4.21 (1.87) | 3.60 (1.83)
  VAS-Physical sedation score | 6.25 (1.50) | 3.69 (1.90) | 3.35 (1.85)
  DIEPSS-Bradykinesia score | 0.25 (0.46) | 0 (0) | 0.10 (0.32)

4. Secondary Outcome: Assessment of Cognitive Functioning-1
Description: CNT(Computerized Neuro-Cognitive Function Test System); The tests included a word fluency test. All of the assessments except the CNT were conducted immediately prior to administration of the medication and at 2 (for risperidone and placebo) or 24 h (for paliperidone ER) after the first and third administrations of the study medications.
  Minimum of Wisconsin card sorting test-Category completed is 0, Maximum is 6, the lower number is worse outcome.
  Minimum of Wisconsin card sorting test-Perseverative response and Trials to complete is 0, Maximum is 128, the lower number is worse outcome.
  Minimum of Wisconsin card sorting test-Perseverative error is 0, Maximum is 128, the higher number is worse outcome.
  Minimum of Word-fluency test is 0 and no maximum value, the higher number is better outcome.
  The score ranges are for subscale score. This outcome measure is reporting a change between baseline and 50hr after third medication.
Time Frame: baseline and 50hr after third medication
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Risperidone | Placebo | Paliperidone ER
Number analyzed (Participants) | 10 | 12 | 10
scores on a scale
  Word-fluency test-Animal | 22.22 (9.46) | 25.42 (4.12) | 23.50 (6.22)
  Word-fluency test-Stationery | 22.56 (7.58) | 26.00 (5.24) | 23.60 (4.70)
  Word-fluency test-"ㄱ" | 17.44 (7.68) | 19.75 (4.54) | 17.10 (5.13)
  Word-fluency test-"ㅅ" | 17.44 (5.85) | 18.25 (4.85) | 16.40 (2.17)
  Word-fluency test-"ㅇ" | 16.11 (4.11) | 17.17 (4.73) | 16.70 (4.27)

5. Secondary Outcome: Symptoms Assessment by Objective Rating Scales
Description: SANS(Scale for the Assessment of Negative Symptoms), NIDSS(Neuroleptic induced Deficit Syndrome Scale) Minimum of NIDSS is -3, maximum of NIDSS is +3. '+' is better outcome, '-' is worse outcome. Minimum of SNAS-Global score is 0, Maximum of SNAS-Global score is 5 The higher number is worse outcome. The zeros are measured and Calcuated value. The score ranges are for subscale score. This outcome measure is reporting a change between baseline and 50hr after third medication.
Time Frame: baseline and 50hr after third medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Placebo | Paliperidone ER
Number analyzed (Participants) | 10 | 12 | 10
units on a scale
  NIDSS-Avolition | -0.85 (0.70) | -0.37 (0.72) | 0.14 (0.78)
  NIDSS-Blunted Affect | -0.70 (0.64) | -0.27 (0.34) | 0.04 (0.67)
  NIDSS-Cognition | -0.66 (0.57) | -0.26 (0.39) | 0.28 (0.61)
  NIDSS-Total | -0.72 (0.59) | -0.29 (0.41) | 0.19 (0.63)
  SANS-Global score for alogia | 0.13 (0.35) | 0 (0) | 0 (0)
  SANS-Global score for blunted affect | 0.25 (0.46) | 0 (0) | 0 (0)

6. Secondary Outcome: Assessment of Cognitive Functioning-2
Description: CNT(Computerized Neuro-Cognitive Function Test System); The tests included the Stroop test, Trail-Making Test B (TMT B). All of the assessments except the CNT were conducted immediately prior to administration of the medication and at 2 (for risperidone and placebo) or 24 h (for paliperidone ER) after the first and third administrations of the study medications Minimum of Stroop test is 0, no maximum limit, the higher number is worse outcome.
  Minimum of Trail making test B is 0 and no maximum limit, the higher number is worse outcome.
  The score ranges are for subscale score. This outcome measure is reporting a change between baseline and 50hr after third medication.
Time Frame: baseline and 50hr after third medication
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Risperidone | Placebo | Paliperidone ER
Number analyzed (Participants) | 10 | 12 | 10
milliseconds
  Stroop test-Color | 15.40 (4.51) | 13.09 (1.67) | 12.68 (1.70)
  Stroop test-Word-color | 21.84 (4.53) | 17.53 (2.97) | 18.31 (3.29)
  Stroop test-Interference score | 6.43 (1.77) | 4.44 (2.01) | 5.63 (2.71)
  Trail making test B | 29.78 (10.24) | 28.42 (7.45) | 31.10 (8.66)

7. Secondary Outcome: Assessment of Cognitive Functioning-3
Description: CNT(Computerized Neuro-Cognitive Function Test System); The tests included Wisconsin Card-Sorting Test (WCST). All of the assessments except the CNT were conducted immediately prior to administration of the medication and at 2 (for risperidone and placebo) or 24 h (for paliperidone ER) after the first and third administrations of the study medications.
  Minimum of Wisconsin card sorting test-Category completed is 0, Maximum is 6, the lower number is worse outcome.
  Minimum of Wisconsin card sorting test-Perseverative response and Trials to complete is 0, Maximum is 128, the lower number is worse outcome.
  Minimum of Wisconsin card sorting test-Trials to complete first category trials is 0, Maximum is 128 and minimum of Wisconsin card sorting test-Perseverative error is 0, Maximum is 128, the higher number is worse outcome.
  The score ranges are for subscale score. This outcome measure is reporting a change between baseline and 50hr after th
Time Frame: baseline and 50hr after third medication
Measure: Mean (Standard Deviation); unit: trials
Arm/Group | Risperidone | Placebo | Paliperidone ER
Number analyzed (Participants) | 10 | 12 | 10
trials
  Wisconsin card sorting test-Category completed | 6.00 (0.00) | 6.00 (0.00) | 6.00 (0.00)
  Wisconsin card sorting test-Perseverative response | 14.11 (6.03) | 13.08 (8.11) | 10.10 (2.96)
  Wisconsin card sorting test-Perseverative error | 10.00 (3.50) | 9.67 (6.11) | 6.50 (1.18)
  WCST-Trials to complete first category trials | 14.00 (7.98) | 11.75 (2.01) | 12.10 (2.42)

ADVERSE EVENTS:
Arm/Group | Risperidone | Placebo | Paliperidone ER
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 5/11 | 2/12 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone (N=11) | Placebo (N=12) | Paliperidone ER (N=11)
Abdominal discomfort(vomiting) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone (N=11) | Placebo (N=12) | Paliperidone ER (N=11)
sedation (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0)
abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The sample size was small, which presents higher risk of a type II error. The time of assessment after administering placebo or risperidone was noon to 2 PM, which may have contributed to the increased reports of sedation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No